CLINICAL TRIAL: NCT00220714
Title: Effectiveness of Long-Acting Risperidone in the Maintenance Treatment of First-Episode Schizophrenia
Brief Title: PREvent First Episode Relapse (PREFER)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIS-SCH-420
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; first-episode; patient compliance; long-acting risperidone; relapse
MeSH Terms: conditions — Schizophrenia; Patient Compliance; Recurrence

INTERVENTIONS:
Drug: atypical antipsychotics:oral vs. long-acting route
Behavioral: Family Psychoeducation

SUMMARY:
Many patients who have recently received a diagnosis of schizophrenia (e.g., "first-episode schizophrenia") respond very well to their antipsychotic medication when they are acutely ill. Once they are more stable, research has shown that first-episode patients need to remain on their antipsychotic medication. Follow-up studies show that stopping medication prematurely is the most common cause of relapse and readmission. It is important to have new ways to help patients stay stable in the community in order for them to continue on with their rehabilitation and recovery process.

Over the last decade, new antipsychotic medications have been developed that are more effective and have fewer side effects than older antipsychotics. The new medicines are often called "atypical", and were only available by pill or capsule for long-term treatment. Most recently, one of the atypical medications - risperidone - became available as a long-acting injection that can be given once every 2 weeks.

The hypothesis of this study is that patients recovering from an acute episode and who then go on to receive a long-acting version of atypical antipsychotic medication (long-acting risperidone microspheres) will stay on their medications for longer than those who take their atypical medication (any available first-line atypical) in the oral (pill) form.

DETAILED DESCRIPTION:
Overview: Before the atypicals were introduced, some of the older antipsychotics were available in oral (pill or capsule) and long-acting (depot) versions. Despite the potential advantages of the depot versions, in those days clinicians in the United States have historically limited the use of long-acting, "depot" antipsychotics to their most treatment-resistant, chronic, patients. Therefore, most clinicians did not routinely consider starting a long-acting antipsychotic early in the course of treatment, such as after the first-episode of schizophrenia.

This whole issue was less relevant after the atypical medications came out, because they were only available in oral versions for long-term treatment. Now that one of the atypical medications (risperidone) is available for use in the United States, the issue of appropriate use of oral vs. long-acting atypical is now very relevant to clinical practice.

For first episode patients, there are been two issues that suggest that the route of medication delivery is an important area to study. First is that almost all first-episode patients will stop their medication too soon. Second, a there now is atypical antipsychotic available in a long-acting preparation (long-acting risperidone, but this option is not often used right away after a first episode, so there is little guidance for clinicians about the effectiveness of long-acting antipsychotics used right away after a first-episode.

Methods: This study compares the effectiveness of the long-acting route of medication to improve adherence and reduce relapse among patients who have been recently diagnosed with schizophrenia or a related psychotic disorder. After patients are stabilized with an atypical antipsychotic and have received patient and family psychoeducation, consenting patients will be randomized to a prospective, random-assignment open-label study comparing any available first-line oral atypical antipsychotic to long-acting risperidone for the maintenance treatment of patients recovering from acute treatment of first-episode schizophrenia.

This study is divided into three study phases. Study Phase I is the acute phase, where consenting patients would be given an acute open-label trial of an oral antipsychotic. Patients who respond within a maximum of 12 weeks to acute therapy will then be invited to participate in Phase II of the study. Patients agreeing to Phase II will then be randomized into staying on their oral antipsychotic medication vs. switching to a long-acting atypical antipsychotic (long-acting risperidone). Patients would be followed for 12 weeks to determine whether or not they accept a recommendation of long-acting antipsychotic or continued oral antipsychotic. Then patients enter into Study Phase III, where they are followed for at the remainder of the year. We want to learn how often patients will accept their doctor's recommendation of a long-acting injection, whether persons taking their antipsychotic medication in long-acting form do better in terms of willingness to stay on their medication, or have better symptom control or fewer side effects, than persons where the doctor recommends the medication in oral (pill) form.

Summary: Patients recently diagnosed as suffering from schizophrenia, e.g. the "first-episode" patient might benefit from an atypical antipsychotic given in a long-acting route of drug- delivery. However, long-acting antipsychotic therapy is not routinely considered in first-episode patients. Studying the acceptance and ultimate effectiveness of a long-acting atypical antipsychotic would be very helpful in understanding how to help patients stay stable and ultimately prevent a revolving door pattern that, if it continues, can be devastating to the recovery process.

ELIGIBILITY:
There is a 2 step inclusion/exclusion criteria, the first being for assessing overall eligibility to be enter, and then, for continued outpatient treatment for schizophrenia when clinically appropriate.

Inclusion criteria for the first phase:

1. Between 16-50 years of age
2. Psychotic symptoms must have persisted at least one month prior to starting the current antipsychotic
3. Continue to show some positive (psychotic) symptoms of schizophrenia
4. A provisional clinical diagnosis of schizophreniform disorder,schizophrenia, or schizoaffective disorder
5. Confirm that there was no previous history of significant pharmacological treatment with an antipsychotic medication
6. Able to fully participate in the informed consent process

Exclusion criteria for Study Phase I

1. Unable to understand informed consent process
2. A history of nonresponse to, or severe adverse events from, any prior exposure to oral risperidone
3. Will not be living close enough to the medical center to return for follow-up visits or assessments
4. Currently receiving medication over objection by court order

Inclusion criteria for Study Phase II

Key criteria for entry into Study Phase II are:

1. Has clinically responded to the oral antipsychotic regimen
2. Willingness to transition to receive evaluation and future pharmacologic treatment at the Schizophrenia Research Service
3. Has retained capacity to understand the risks and benefits of the maintenance treatment with antipsychotics
4. Willingness to sign informed consent to go into Study Phase II

Exclusion criteria for Study Phase II

1. Has not responded to the current oral antipsychotic regimen, or has had significant side effects to oral risperidone
2. Explicit refusal to even consider the possibility of receiving maintenance antipsychotic by long-acting injection

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80
Dates: Start 2004-11; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Likelihood of accepting a recommendation of long-acting atypical antipsychotic medication
Compare the time until the first episode of antipsychotic nonadherence as defined by 2 or more weeks of continuous and intentional cessation of all prescribed antipsychotic medication
Compare the total amount of outpatient days spent adherent to antipsychotic medication as a proportion of outpatient days in the study
Compare patient and family attitudes and satisfaction with antipsychotic medication given by long-acting route vs. oral route of drug delivery
5. Modify and adapt psychoeducational material designed for multiple episode patients to better fit the needs of recently diagnosed patients with schizophrenia.

SECONDARY OUTCOMES:
Compare the likelihood of relapse and rehospitalization between long-acting atypical antipsychotic with all available first-line oral atypical agents
Compare the longitudinal course of symptoms and side effects of those remaining on long-acting atypicals to those remaining on oral antipsychotic regimens
Compare outcome differences between intent-to-treat assignments with actual observed treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Weiden, M.D., Principal Investigator — State University of New York - Downstate Medical Center
Locations (2):
- United States (2):
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York

REFERENCES:
- [Derived] Weiden PJ, Schooler NR, Weedon JC, Elmouchtari A, Sunakawa-McMillan A. Maintenance treatment with long-acting injectable risperidone in first-episode schizophrenia: a randomized effectiveness study. J Clin Psychiatry. 2012 Sep;73(9):1224-33. doi: 10.4088/JCP.11m06905. Epub 2012 Aug 7. PMID 22938760
- [Derived] Weiden PJ, Schooler NR, Weedon JC, Elmouchtari A, Sunakawa A, Goldfinger SM. A randomized controlled trial of long-acting injectable risperidone vs continuation on oral atypical antipsychotics for first-episode schizophrenia patients: initial adherence outcome. J Clin Psychiatry. 2009 Oct;70(10):1397-406. doi: 10.4088/JCP.09m05284yel. PMID 19906343